CLINICAL TRIAL: NCT06339918
Title: Combined Effects of Kegel Exercises and 4-7-8 Breathing Technique on Pain Intensity, Symptom Severity and Functional Activity in Primary Dysmenorrhea
Brief Title: Combined Effects of Kegel Exercises and 4-7-8 Breathing Technique in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0570
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Primary Dysmenorrhea
Keywords: Kegel Exercises; Breathing Exercises; Relaxation Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel Exercise with4-7-8 Breathing technique group: (Experimental): GroupAwill be given the intervention of kegel exercises as well as 4-7-8 breathing techniques for about 15 minutes per session for a total of 8 weeks with 4 sessions per week. To perform kegel exercises, tighten pelvic floor muscles like trying to hold in urine and stool. 4-7-8 breathing Technique can be performed by telling the participant to inhale to the count of 4. Hold their breath for 7 counts. To the count of 8, release air via their mouth.
  Interventions: Other: KegelExercise; Other: 4-7-8 breathing technique
- 4-7-8 Breathing Technique group (Active Comparator): In this group, we only perform the 4-7-8 Breathing Technique by telling the participant to inhale to the count of 4. Hold their breath for 7 counts. To the count of 8, release air via their mouth.
  Interventions: Other: 4-7-8 breathing technique

INTERVENTIONS:
Other: KegelExercise — Kegel exercises (also called pelvic floor exercises)will be used to strengthen the pelvic floor muscles it will involve repeatedly contracting and relaxing the muscles that form part of the pelvic floor.
  Arms: Kegel Exercise with4-7-8 Breathing technique group:
Other: 4-7-8 breathing technique — This can be performed in the following way: Participants taking part should locate a comfy spot to sit. Inhale to the count of 4. Hold their breath for 7 counts. To the count of 8, release air via their mouth.

SUMMARY:
A randomized clinical trial will be conducted at Riphah International University QIE Campus in Lahore, using non-probability convenience sampling with 28 participants. Criteria include women aged 14-26, nulliparous, experiencing primary dysmenorrhea, with normal menstrual cycles and the ability to exercise independently. Group A will receive kegel exercises and 4-7-8 breathing techniques over 8 weeks, while Group B will only receive the breathing technique. Assessments will be done on menstrual cycle days, with follow-ups at weeks 4 and 8 using specific scales. Data will be analyzed using SPSS version 27.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial. Riphah International University QIE Campus in Lahore will serve as the site of data collecting and intervention services. Non-probability convenience sampling will be the method of sampling. The study's sample size will be 28 participants. Inclusion criteria for this study will be: women between ages 14-26 years, nulliparous women, with a score greater than 4 in WALIDD primary dysmenorrhea intensity scales, history of normal menstrual cycles that lasts 3-7 days and ranged from 21- 35 days, ability to perform exercises independently. Group A will be given kegel exercises as well as 4-7-8 breathing techniques for a total of 8 weeks with 4 sessions per week. Whereas, group B will be given the 4-7-8 breathing technique only. Initial assessment will be taken on the 3rd day of menstrual period. Follow-up assessment will be taken after week 4 post interventions and final assessment will be done after week 8 post intervention. WaLIDD primary dysmenorrhea intensity scale, Pain Self-Efficacy Questionnaire (PESQ), and Numeric Pain Rating Scale (NPRS) will be the data collecting instruments.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Women with a score greater than 4 on WALIDD primary dysmenorrhea intensity scale
* Women having a history of normal menstrual cycles that lasts 3-7 days and range from 21- 35 days.
* Ability to perform exercises independently

Exclusion Criteria:

* Women with very mild primary dysmenorrhea
* Women treated for ovarian cysts or other gynecological issues
* Women currently taking medication for dysmenorrhea
* History of any systemic illness
* A history of psychological conditions that could influence the perception of pain and functional activity.

Ages: 14 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | up to 8 weeks
  TheNPRSisa popular patient-reported response scale is the NPRS. The most widely used form of the NPRS is the ordinal 11-point version (0-no pain, 10-most extreme pain). A line or bar that is horizontal is the standard format. The NPRS is anchored by phrases that describe extremes of pain severity.
WALIDD Primary Dysmenorrhea Intensity Scale | up to 8 weeks
  WaLIDD stands for working ability, location, intensity, days of pain, dysmenorrhea. It is used to diagnose Primary dysmenorrhea as well its pain intensity and severity of symptoms. It is a new tool established and used in many researches and practices as a questionnaire to evaluate whether women are suffering from primary dysmenorrhea or not. The WaLIDD instrument is part of a confidential questionnaire that inquires about every factor to be examined, as well as details about age, menarche, menstrual cycle features, type and number of nonsurgical treatments used to manage dysmenorrhea, number of days of medical leave taken for dysmenorrhea.
Pain Self-Efficacy Questionnaire (PSEQ) | up to 8 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a valid instrument that is widely used to evaluate a person's comfort level with chronic pain management. Rhe PSEQ measures self-efficacy beliefs in pain management and how important it is to comprehend how pain affects both functional and emotional elements of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal Zahid, MS*, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Riphah International University Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abreu-Sanchez A, Parra-Fernandez ML, Onieva-Zafra MD, Ramos-Pichardo JD, Fernandez-Martinez E. Type of Dysmenorrhea, Menstrual Characteristics and Symptoms in Nursing Students in Southern Spain. Healthcare (Basel). 2020 Aug 26;8(3):302. doi: 10.3390/healthcare8030302. PMID 32858887
- [Background] Bernardi M, Lazzeri L, Perelli F, Reis FM, Petraglia F. Dysmenorrhea and related disorders. F1000Res. 2017 Sep 5;6:1645. doi: 10.12688/f1000research.11682.1. eCollection 2017. PMID 28944048
- [Background] Bakhsh H, Algenaimi E, Aldhuwayhi R, AboWadaan M. Prevalence of dysmenorrhea among reproductive age group in Saudi Women. BMC Womens Health. 2022 Mar 19;22(1):78. doi: 10.1186/s12905-022-01654-9. PMID 35305636
- [Background] Matsas A, Sachinidis A, Lamprinou M, Stamoula E, Christopoulos P. Vitamin Effects in Primary Dysmenorrhea. Life (Basel). 2023 Jun 1;13(6):1308. doi: 10.3390/life13061308. PMID 37374091